CLINICAL TRIAL: NCT01149356
Title: A Phase I Dose Escalation Trial of RO4929097 Administered in Combination With Exemestane in Pre- and Postmenopausal Patients With ER + Metastatic Breast Cancer
Brief Title: RO4929097 And Exemestane in Treating Pre- and Postmenopausal Patients With Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Manufacturer discontinued drug development.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2010-02181; NCI-2010-02181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC-8539; CDR0000675612; 8539 (Other: Moffitt Cancer Center); 8539 (Other: CTEP); N01CM00100 (NIH); P30CA076292 (NIH)
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Estrogen Receptor Positive; HER2/Neu Negative; Male Breast Carcinoma; Recurrent Breast Carcinoma; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — exemestane; 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Goserelin

ARMS (2):
- Arm I (Experimental): Patients receive oral exemestane once daily on days 1-21 and oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Exemestane; Drug: Gamma-Secretase Inhibitor RO4929097; Drug: Goserelin Acetate
- Arm II (Active Comparator): Patients receive exemestane as in arm I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Exemestane; Drug: Goserelin Acetate

INTERVENTIONS:
Drug: Exemestane — Given orally
  Other Names: Aromasin; FCE-24304
Drug: Gamma-Secretase Inhibitor RO4929097 — Given orally
  Other Names: RO4929097
  Arms: Arm I
Drug: Goserelin Acetate — Given subcutaneously to premenopausal patients
  Other Names: ZDX; Zoladex

SUMMARY:
This partially randomized phase I trial is studying the side effects and the best dose of RO4929097 when given together with exemestane and to see how well it works compared to exemestane alone in treating premenopausal and postmenopausal patients with advanced or metastatic breast cancer. Estrogen can cause the growth of breast cancer cells. Hormone therapy using exemestane may fight breast cancer by lowering the amount of estrogen the body makes. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving exemestane together with RO4929097 may kill more breast cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum-tolerated dose of gamma-secretase inhibitor RO4929097 (RO4929097) in combination with exemestane in pre- and postmenopausal patients with estrogen receptor-positive (ER+) advanced or metastatic breast cancer.

II. Determine the safety and tolerability of this regimen in these patients. III. Determine the progression-free survival of patients treated with exemestane with vs without RO4929097.

SECONDARY OBJECTIVES:

I. Determine the overall tumor response rate in patients treated with these regimens.

II. Determine the overall survival of patients treated with these regimens. III. Determine the safety of these regimens in these patients. IV. Determine the quality of life of patients treated with these regimens. V. Identify biomarkers of response to treatment or toxicity.

OUTLINE: This is a multicenter, phase I, dose-escalation study of gamma-secretase inhibitor RO4929097.

Patients receive oral exemestane once daily on days 1-21 and oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are stratified according to menopausal status (pre- vs postmenopausal) and visceral disease (yes vs no). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive exemestane as in phase I and oral gamma-secretase inhibitor RO4929097 at the MTD determined in phase I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive exemestane as in arm I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

In addition to exemestane, pre-menopausal patients receive goserelin subcutaneously every 28 days. Patients may undergo blood and tissue sample collection for correlative studies.

Patients may complete quality-of-life questionnaires at baseline and periodically during study using the Functional Assessment of Cancer Therapy for Breast Cancer (FACT-B).

After completion of study therapy, patients are followed up for 4 weeks and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer

  * Locally advanced or metastatic disease for which curative measures are not effective

    * Relapsed disease with (or within 6 months of discontinuation of) an adjuvant nonsteroidal aromatase inhibitor or tamoxifen
    * Progressive disease during treatment with first- or second-line hormonal therapy that could include a nonsteroidal aromatase inhibitor, tamoxifen, or fulvestrant
  * Recurrent disease

    * No locally recurrent resectable disease
  * Histologically confirmed estrogen receptor-positive (ER+) by IHC

    * Must have ≥ 5% strong staining for ER+ or ≥ 10% weak staining
* Measurable disease defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques OR as ≥ 10 mm by spiral CT scan
* No HER2/neu-positive disease
* No known brain metastases
* Pre- or postmenopausal status
* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* WBC ≥ 3,500/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 2 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Able to swallow and retain oral medication
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for ≥ 12 months after completion of study therapy
* More than 5 years since other invasive cancer except basal or squamous cell cancer of the skin or cervical carcinoma in situ
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gamma-secretase inhibitor RO4929097 or other agents used in the study
* No history of torsades de pointes
* No malabsorption syndrome or other condition that would interfere with intestinal absorption (e.g., ulcerative colitis)
* Not serologically positive for hepatitis B or C, have a history of liver disease, other forms of hepatitis, or cirrhosis
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection requiring parenteral antibiotics
  * Impairment of lung function (e.g., chronic obstructive pulmonary disease or lung conditions requiring oxygen therapy)
  * Symptomatic congestive heart failure (NYHA class III-IV heart disease)
  * Unstable angina pectoris, angioplasty, stenting, and or myocardial infarction within the past 6 months
  * Uncontrolled hypertension (systolic BP > 180 mm Hg or diastolic BP > 100 mm Hg on 2 consecutive measurements separated by a 1-week period) despite adequate medical support
  * Clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, torsades de pointes, ventricular tachycardia that is symptomatic, or requiring treatment)
  * A requirement for antiarrthymics or other medications known to prolong QTC
  * Uncontrolled diabetes (hyperosmolar state, ketoacidosis, etc.)
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* No baseline QTcF > 450 msec (male) or > 470 msec (female)
* See Disease Characteristics
* Fully recovered from all previous adverse events
* No prior exemestane for metastatic or recurrent breast cancer, or within the past 6 months in the adjuvant setting
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* At least 2 weeks since prior radiotherapy
* At least 2 weeks since prior and no other concurrent investigational agents
* No prior exposure to γ-secretase inhibitors
* No concurrent medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®)
* No other concurrent CYP3A4 substrates, inducers, or inhibitors
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies, including chemotherapy, radiotherapy, surgery, immunotherapy, hormonal therapy, or biologic therapy
* No concurrent medications or food that may interfere with the metabolism of gamma-secretase inhibitor RO4929097, including ketoconazole and grapefruit juice
* No concurrent antiarrhythmics or other medications known to prolong QTc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) based on CTCAE version 3 grade | Up to 70 days
  Will be summarized by body system, preferred term, verbatim of adverse event, intensity, and relationship to each study drug (BMS-936558 and/or the peptide vaccine).
Time to relapse | Up to 2 years
  Time to relapse will be summarized using descriptive statistics.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Julie Means-Powell, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee